CLINICAL TRIAL: NCT03469648
Title: Incidence of Intraoperative Positive Air-Test
Brief Title: Intraoperative Air-Test
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Carlos Ferrando, Anesthesiologist, Fundación para la Investigación del Hospital Clínico de Valencia
Other Study IDs: Air-Test
Record Dates: First submitted 2018-03-07; First posted 2018-03-19 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Patients With ASA Status I-III Scheduled for Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Air-Test — The Air Test simply consisted in breathing room air for 5 min during anesthesia while measuring peripheral oxygen saturation by Pulse oximetry

SUMMARY:
Although imaging techniques are the reference standard to diagnose alveolar collapse, in the postoperative period and using the peripheral hemoglobin oxygen saturation (SpO2), a non-invasive simple and accurate test (Air-Test) was recently validated to diagnose alveolar collapse.

The aim of this study is to non-invasively describe the incidence of intraoperative atelectasis with the Air-Test in an unselected surgical population. In addition, we attempt to describe the association between positive Air-Test and the patient´s preoperative or intraoperative variables.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) I-IV
* General Anesthesia
* Mechanical ventilation

Exclusion Criteria:

* age < 18 years old
* pregnancy
* patients undergoing cardiothoracic surgery
* ASA physical status V

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included consecutive patients who were scheduled for surgery with general anesthesia and mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Patients with positive Air-Test | During surgery
  Positive Air-Test defined as SpO2 < 97% while breathing room air

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Carlos Ferrando, Valencia
  - Department of Anesthesia and Critical Care; Hospital Clinico Universitario, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrando C, Tusman G, Suarez-Sipmann F, Leon I, Pozo N, Carbonell J, Puig J, Pastor E, Gracia E, Gutierrez A, Aguilar G, Belda FJ, Soro M. Individualized lung recruitment maneuver guided by pulse-oximetry in anesthetized patients undergoing laparoscopy: a feasibility study. Acta Anaesthesiol Scand. 2018 May;62(5):608-619. doi: 10.1111/aas.13082. Epub 2018 Jan 29. PMID 29377061
- [Background] Ferrando C, Romero C, Tusman G, Suarez-Sipmann F, Canet J, Dosda R, Valls P, Villena A, Serralta F, Jurado A, Carrizo J, Navarro J, Parrilla C, Romero JE, Pozo N, Soro M, Villar J, Belda FJ. The accuracy of postoperative, non-invasive Air-Test to diagnose atelectasis in healthy patients after surgery: a prospective, diagnostic pilot study. BMJ Open. 2017 May 29;7(5):e015560. doi: 10.1136/bmjopen-2016-015560. PMID 28554935